CLINICAL TRIAL: NCT06426004
Title: Community Interventions to Address Health Disparities in the Care of Normal Pressure Hydrocephalus (NPH) in Maryland
Brief Title: Addressing Health Disparities in Normal Pressure Hydrocephalus (NPH) in Maryland
Acronym: NPH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: IRB00028028
Record Dates: First submitted 2024-05-15; First posted 2024-05-23 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Normal Pressure Hydrocephalus; Hakim Syndrome
MeSH Terms: conditions — Hydrocephalus, Normal Pressure | interventions — Physicians, Primary Care

STUDY DESIGN:
Intervention Model Description: The investigators will develop three layers of interventions that involve educational elements about NPH and evaluate which provides the most benefit including referrals to NPH related care. 1) Patients identified from the first part of the study with possible NPH symptoms will receive intervention 2) Patients, and the Primary Care Providers (PCPs) receive intervention, and 3) patients, and PCP receive intervention and with additional community health workers (CHWs) assisting providers with managing the patient care including referrals, addressing socioeconomic barriers, transportation to receive care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients and the patient's family (Experimental): All patients and the patient's family will receive NPH-related education.
  Interventions: Other: patients will receive NPH education; Other: primary care physicians (PCPs) will receive professional NPH education; Other: A community health worker will assist PCP
- PCPs Training (Experimental): Primary Care Provider (PCP) will receive NPH education.
  Interventions: Other: primary care physicians (PCPs) will receive professional NPH education; Other: A community health worker will assist PCP
- CHWs assist PCPs (Experimental): A community health worker (CHW) will assist PCP.
  Interventions: Other: A community health worker will assist PCP

INTERVENTIONS:
Other: patients will receive NPH education — Patients will benefit from the Hydrocephalus Association's (HA) educational strategy for idiopathic normal pressure hydrocephalus (iNPH) emphasizes patient collaboration in the development of educational materials specifically for this condition. HA has a library of assets that include PowerPoint presentations, videos, and online and print educational materials. There will be also in-person outreach resulting recruitment, website (the study website and HA website), webform (with a symptom of gait, dementia, and bladder symptoms), YouTube videos. The investigators will also go to the communities like senior centers, health fair, and churches, then we will give a talk about iNPH. These resources will be carefully adjusted to suit low-income demographics, guided by feedback from Baltimore audiences and HA's iNPH volunteers.
  Arms: Patients and the patient's family
Other: primary care physicians (PCPs) will receive professional NPH education — A comprehensive professional development program for PCPs and CHWs, featuring presentations, educational videos, webinars, and tools on iNPH diagnosis, treatment, and care management. Provider Continuing Medical Education (CME) credits will be offered for in-person lectures, aiming to equip PCPs with the skills needed to address iNPH in low-income settings effectively
  Arms: PCPs Training; Patients and the patient's family
Other: A community health worker will assist PCP — A community health worker will assist PCP to identify barriers and help overcome these barriers in order for patient to access iNPH care.

SUMMARY:
The study aims to estimate Normal Pressure Hydrocephalus (NPH) prevalence and evaluate health equity gaps in Baltimore and Maryland based on zip codes and race, with a focus on the Black community. Interventions will include educational elements about NPH and three layers targeting patients, Primary Care Providers, and community health workers to enhance care access. Short-term outcomes will measure referrals to specialists, while long-term outcomes will assess healthcare utilization. The study aims to identify and reduce racial disparities in NPH care access, informing intervention strategies for NPH and other surgical areas.

DETAILED DESCRIPTION:
This proposal responds to an established need for developing an evidence-based and community-informed approach to address health disparities in specialty surgical clinics where barriers to accessing care are multiplied along each level of the referral pathway. The study will focus on Normal Pressure Hydrocephalus (NPH) related care - a clinical syndrome characterized excess cerebrospinal fluid (CSF) in the brain resulting in symptoms of falls, dementia, and urinary incontinence, that is treated surgically by shunting to remove excess fluid from the brain. This disorder afflicts an estimated about 750,000 Americans, and prevalence increases with age. Limited information regarding racial and socioeconomic contributing factors associated with diagnosis and treatment is available.

Studies show NPH goes underdiagnosed in the USA. In the first part of the study the investigators will estimate NPH prevalence, the health equity gap in Baltimore and greater Maryland (MD), the health equity gap based on Zip Code as a marker of sociodemographic community status, and the health equity gap based on race, looking at the Black community, which comprises over 60% of the Baltimore and 30% in MD population. In the second part of the study, the investigators will develop three layers of interventions that involve educational elements about NPH and evaluate which provides the most benefit including referrals to NPH related care. 1) Patients identified from the first part of the study with possible NPH symptoms will receive intervention 2) Patients, and the Primary Care Providers (PCPs) receive intervention, and 3) patients, and PCP receive intervention and with additional community health workers (CHWs) assisting providers with managing the patient care including referrals, addressing socioeconomic barriers, transportation to receive care.

The success of these interventions will be evaluated by short-term outcomes such as referrals to specialists including neurologists and neurosurgeons every 6 months, and long-term outcomes such as healthcare utilization including screening for shunt surgery within 12 months. This study aims to identify racial disparities in access to NPH care and intervention outcomes will evaluate the effect of different interventions on reducing racial disparities and to help developing a referral system to address the needs of most vulnerable population and Zip Codes in Baltimore and greater MD. Using the results of this study will help to identify gaps, understand the best intervention, and develop intervention strategies not only for NPH but potentially other surgical areas.

ELIGIBILITY:
Inclusion Criteria:

* People over 65 years old who have completed the Annual Wellness Survey (AWV) survey
* have a clinical profile in the Hopkins Epic data sets
* live in Maryland

Exclusion Criteria:

* People under 65 years old will be excluded if they have not completed the AWV survey
* do not live in Maryland

Community Health Worker (CHW) Inclusion Criteria:

* certified Community Health Workers from Maryland
* completed accredited training by the Maryland Department of Health

Primary Care Physician inclusion criteria:

* must have patients in Johns Hopkins University AWV

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
number of referrals | 6 months
  number of referrals for suspicion of NPH to neurologists or neurosurgeons
number of screenings | 12 months
  number of screenings for shunt surgery
number of screenings | 24 months
  number of screenings for shunt surgery

SECONDARY OUTCOMES:
number of NPH's consultations | 24 months
  number of patients who have received a consultation

OTHER OUTCOMES:
number of referrals | 12 months and 24 months
  referrals for physical therapy, occupational therapy, psychiatry, neurology - movement disorder specialist, neurology neuropathy specialist, orthopedic surgery, neurosurgery- spine specialist, neuropsychologist

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Zare, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (2):
- United States (2):
  - Johns Hopkins University and Hospital, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and analytic plan will be freely available. In addition to analytical files, the Stata, Statistical Analysis System (SAS), R codes and programs and data dictionary will be available to researchers approved by one of the study's Principal Investigators to receive data. All papers must include an acknowledgment section that includes the funding source.
Supporting Information: SAP, CSR
Time Frame: The investigators will release the data 2 years after finishing up the study on April 2030.